CLINICAL TRIAL: NCT02244775
Title: Use of Avanta Metacarpophalangeal (MCP) Joint Implant Finger Prosthesis, Humanitarian Use Device
Status: Approved for marketing | Type: Expanded Access
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-090
Record Dates: First submitted 2014-09-12; First posted 2014-09-19 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Arthroplasty of the MCP Joint
Keywords: osteo-arthritis; post traumatic arthritis

INTERVENTIONS:
Device: SR™MCP

SUMMARY:
The purpose of this study is to allow patients to undergo surgery with the SR™ MCP (Metacarpophalangeal) Implants for finger arthritis. This is NOT a research study, but rather, a requirement by the FDA for humanitarian use of device.

DETAILED DESCRIPTION:
The purpose of this IRB approved study is to allow patients to undergo surgery with the SR™ MCP (Metacarpophalangeal) Implants. This is NOT a research study, but rather, a requirement by the FDA for humanitarian use of device. Use of the SR™ MCP is approved for humanitarian use by the FDA when either the patient is in need of a revision of failed MCP prothesis(es) or the patient expects to place his/her hand under loading situation which preclude the use of an alternative implant in the painful osteo-arthritic and post traumatic arthritic MCP joint.

ELIGIBILITY:
Inclusion Criteria:

* patient is in need of a revision of failed MCP prosthesis(es)
* patient expects to place his/her hands under loading situations which preclude the use of an alternative implant in the painful osteo-arthritic and post traumatic arthritic MCP joint

Exclusion Criteria:

* patient is not in need of a revision of a failed MCP prothesis(es)
* patient is eligible to use an alternative implant

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital for Special Surgery, New York, New York, United States